CLINICAL TRIAL: NCT04883541
Title: Assistant Professor,Faculty of Health Sciences Department of Midwifery, Uskudar University, Istanbul, Turkey
Brief Title: Effects of Yoga and Meditation on The Birth Process
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Collaborators: Biruni University (Other)
Responsible Party: Principal Investigator, Tuğba YILMAZ ESENCAN, Assistant Professor, Uskudar University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: Uskudar
Record Dates: First submitted 2021-04-17; First posted 2021-05-12 (Actual); Results first posted 2021-08-09 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Birth, First; Labor Pain; State Anxiety; Self Efficacy
Keywords: Labour Preparation Class; Labour Support; Meditation; Pregnancy Yoga
MeSH Terms: conditions — Labor Pain; Anxiety Disorders | interventions — Yoga; Meditation

STUDY DESIGN:
Intervention Model Description: The present study was conducted as a randomized controlled study.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: For Randomization, when the experiment and control group were created, support was received from pregnancy school instructors and groups, and pregnant women were determined by using the method of envelope selection. Pregnancy school instructors asked the group volunteering to participate in the study to independently choose one of two blue or red colored envelopes. Those who chose the blue envelope formed the experiment group, and those that chose the red envelope were taken into the control group. The envelope selection process continued until the desired numbers were reached. The researcher was told advised of the groups to which subjects were included by the pregnancy school instructor only after the subjects were chosen.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Study Group (Experimental): Pregnant women participated in the applications, which lasted two days a week, for ten weeks, and for 60 minutes a day.
  Interventions: Behavioral: yoga and meditation
- Control Group (Placebo Comparator): The control group was only given delivery preparation training for 6 weeks, and the birth processes were followed by routine follow-ups.
  Interventions: Behavioral: Birth preparation training

INTERVENTIONS:
Behavioral: yoga and meditation — The pregnant women in the study group were given yoga and meditation classes, which included a total of twenty 10-week lessons, which were done by the researchers as 6-week birth preparation training, and with the onset of the birth action, birth processes were followed in the course of labour period yoga and meditation.
  Arms: The Study Group
Behavioral: Birth preparation training — The control group was only given delivery preparation training for 6 weeks, and the birth processes were followed by routine follow-ups.
  Arms: Control Group

SUMMARY:
Introduction: Today it is seen that women lose their birthing strength, give the control to healthcare personnel during labour and the rate of c-section or interventional labour is increasing. For this reason, the importance of yoga, meditation and breath awareness practices increases during pregnancy and birth. The study was carried out as a randomized control trial with the purpose of examining the impact of yoga and meditation during pregnancy and labour on the labour process.

Methods: The study was completed with 90 primiparous pregnant women in total, 30 in experimental group and 60 in control group. The data was collected using State Trait Anxiety Inventory, Wijma Delivery Expectancy/Experience Questionnaire A, The Childbirth Self-Efficacy Scale Short Form, Wijma Delivery Expectancy/Experience Questionnaire Version B and Visual Analogue Scale. Pregnant women in experimental group did yoga and meditation for 60 minutes 2 times a week for 10 weeks. Innatal period yoga and meditation practices were continued in experimental group during labour.

DETAILED DESCRIPTION:
METHODS

Study design:

The present study was conducted as a randomized controlled study. The study was conducted on pregnant women who applied to the pregnancy school of an educational and research hospital on the Anatolian side of Istanbul province between October 2016 and May 2018, and who met the criteria for acceptance of the study.

Setting and samples:

All pregnant women attending the pregnancy school, who agreed to participate in the research, and met the research conditions within the study dates constituted the research population. The sampling of the study was created with the simple random method as the experiment and control group with individuals who met the criteria of the study and who were accepted to participate. In this respect, pregnant women, who were primiparous and between 20-36 gestational weeks, who had single fetuses, expected to give birth normally and spontaneously, with no pregnancy complications and systemic disease, and who could speak Turkish, were included in the study. Power Analysis was made by using the G*Power (v3.1.7) Program to determine the sampling number of the study. According to Cohen's effect size coefficients and other calculations, it was assumed that the evaluations between the two independent groups would have a large impact size (d=0.50). It was also decided that there should be at least 26 people in the groups, and considering that there might be losses in the study process, 30 people were included in the experimental group, and 60 people in the control group, making 90 people in total.

For Randomization, when the experiment and control group were created, support was received from pregnancy school instructors and groups, and pregnant women were determined by using the method of envelope selection. Pregnancy school instructors asked the group volunteering to participate in the study to independently choose one of two blue or red colored envelopes. Those who chose the blue envelope formed the experiment group, and those that chose the red envelope were taken into the control group. The envelope selection process continued until the desired numbers were reached. The researcher was told advised of the groups to which subjects were included by the pregnancy school instructor only after the subjects were chosen.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women,
* Primiparous and between 20-36 gestational weeks,
* Single fetuses, expected to give birth normally and spontaneously,
* No pregnancy complications and systemic disease,
* Speak Turkish

Exclusion Criteria:

* Being unable to speak Turkish
* Having a history of serious illness that threatens life or because of these reasons.
* Currently or previously due to a serious mental weakness or illness
* Being diagnosed with a psychiatric diagnosis and being treated for this reason,
* Being multiparous,
* Multiple pregnancies, being in the gestational week less than 20 weeks and greater than 36 weeks,
* Having a diagnosis that constitutes an obstacle to physical activity

Ages: 21 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women
Enrollment: 153 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-01-01 (Actual); Study Completion 2018-01-30 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: starting 6 months after publication
Access Criteria: JOURNAL EDITOR AND REFEREES TO BE PUBLISHED

REFERENCES:
- [Background] Dick-Read G. Childbirth Without Fear: The Principles and Practice of Natural Childbirth. Second edition. UK: Pinter & Martin Ltd; 2013. 56-100.
- [Background] Rathfisch G. Natural Philosophy of Birth. Istanbul: Nobel Medical Bookstores; 2012.
- [Background] Öner N, LeCompte A. State Trait Anxiety Inventory Handbook, Istanbul; Boğaziçi University Publications;1983.
- [Background] Lecompte A, Öner N. A study on the adaptation and standardization of the state-trait anxiety inventory to Turkish. IX. National Psychiatry and Neurological Sciences Congress Studies 1975;457-462.
- [Background] Erkaya R, Karabulutlu Ö, Çalıka YK. Defining childbirth fear and anxiety levels in pregnant women procedia. Social and Behavioral Sciences 2017; 237:1045-1052.
- [Background] Gönenç İM, Çakırer-Çalbayram N. Contributions of pregnancy school program, opinions of women on the education and their post-education experiences. Journal of Human Sciences 2017; 14(2), 1609-1620. doi:10.14687/jhs.v14i2.4424.
- [Background] Çiçek Ö, Okumuş H. Doğumda öz-yeterlilik algisi: önemi ve etkileyen faktörler, Self-Efficacy perception at birth: its importance and effective factors. International Refereed Journal Ofgynaecological Diseases And Maternal Child Health 2017; 35-49.
- [Background] Greathouse, K. The Nightmare of childbirth: the prevalence and predominant predictor variables for tokophobia in American women of childbearing age [PhD dissertation],. The School of Professional Psychology, Chicago; 2014.
- [Background] Maharana S, Nagarathna R, Padmalatha V, Nagendra HR, Hankey A. The Effect of Integrated Yoga on Labor Outcome: A Randomized Controlled Study. International Journal of Childbirth 2013;(3):165-77. DOI: 10.1891 / 2156-5287.3.3.165.
- [Background] Karakuş A, Şahin NH. The attitudes of women toward mode delivery after childbirth. International Journal of Nursing and Midwifery 2011; 3(5): 60-65. https://doi.org/10.5897/IJNM.9000042.
- [Background] Salomonsson B. Fear is in the air : Midwives´ perspectives of fear of childbirth and childbirth self-efficacy and fear of childbirth in nulliparous pregnant women [PhD dissertation], Linköping University Medical Dissertations, Sweden, 2012; ISBN 978-91-7519-780-7 ISSN 0345-0082.
- [Result] Sercekus P, Baskale H. Effects of antenatal education on fear of childbirth, maternal self-efficacy and parental attachment. Midwifery. 2016 Mar;34:166-172. doi: 10.1016/j.midw.2015.11.016. Epub 2015 Nov 27. PMID 26656473
- [Result] Simkin P, Bolding A. Update on nonpharmacologic approaches to relieve labor pain and prevent suffering. J Midwifery Womens Health. 2004 Nov-Dec;49(6):489-504. doi: 10.1016/j.jmwh.2004.07.007. PMID 15544978
- [Result] Steel A, Adams J, Sibbritt D, Broom A, Frawley J, Gallois C. Relationship between complementary and alternative medicine use and incidence of adverse birth outcomes: an examination of a nationally representative sample of 1835 Australian women. Midwifery. 2014 Dec;30(12):1157-65. doi: 10.1016/j.midw.2014.03.015. Epub 2014 Mar 29. PMID 24742636
- [Result] Polis RL, Gussman D, Kuo YH. Yoga in Pregnancy: An Examination of Maternal and Fetal Responses to 26 Yoga Postures. Obstet Gynecol. 2015 Dec;126(6):1237-1241. doi: 10.1097/AOG.0000000000001137. PMID 26551176
- [Result] Wijma K, Wijma B, Zar M. Psychometric aspects of the W-DEQ; a new questionnaire for the measurement of fear of childbirth. J Psychosom Obstet Gynaecol. 1998 Jun;19(2):84-97. doi: 10.3109/01674829809048501. PMID 9638601
- [Result] Korukcu O, Kukulu K, Firat MZ. The reliability and validity of the Turkish version of the Wijma Delivery Expectancy/Experience Questionnaire (W-DEQ) with pregnant women. J Psychiatr Ment Health Nurs. 2012 Apr;19(3):193-202. doi: 10.1111/j.1365-2850.2011.01694.x. Epub 2012 Jan 20. PMID 22260727
- [Result] Lowe NK. Maternal confidence for labor: development of the Childbirth Self-Efficacy Inventory. Res Nurs Health. 1993 Apr;16(2):141-9. doi: 10.1002/nur.4770160209. PMID 8502766
- [Result] Ip WY, Chan D, Chien WT. Chinese version of the Childbirth Self-efficacy Inventory. J Adv Nurs. 2005 Sep;51(6):625-33. doi: 10.1111/j.1365-2648.2005.03548.x. PMID 16129013
- [Result] Korukcu O, Bulut O, Kukulu K. Psychometric Evaluation of the Wijma Delivery Expectancy/Experience Questionnaire Version B. Health Care Women Int. 2016;37(5):550-67. doi: 10.1080/07399332.2014.943838. Epub 2014 Oct 8. PMID 25119342
- [Result] Wewers ME, Lowe NK. A critical review of visual analogue scales in the measurement of clinical phenomena. Res Nurs Health. 1990 Aug;13(4):227-36. doi: 10.1002/nur.4770130405. PMID 2197679
- [Result] Stoll K, Edmonds JK, Hall WA. Fear of Childbirth and Preference for Cesarean Delivery Among Young American Women Before Childbirth: A Survey Study. Birth. 2015 Sep;42(3):270-6. doi: 10.1111/birt.12178. Epub 2015 Jun 24. PMID 26104997
- [Result] Sydsjo G, Blomberg M, Palmquist S, Angerbjorn L, Bladh M, Josefsson A. Effects of continuous midwifery labour support for women with severe fear of childbirth. BMC Pregnancy Childbirth. 2015 May 15;15:115. doi: 10.1186/s12884-015-0548-6. PMID 25976219
- [Result] Campbell VR, Nolan M. A qualitative study exploring how the aims, language and actions of yoga for pregnancy teachers may impact upon women's self-efficacy for labour and birth. Women Birth. 2016 Feb;29(1):3-11. doi: 10.1016/j.wombi.2015.04.007. Epub 2015 May 29. PMID 26028282
- [Result] Salomonsson B, Gullberg MT, Alehagen S, Wijma K. Self-efficacy beliefs and fear of childbirth in nulliparous women. J Psychosom Obstet Gynaecol. 2013 Sep;34(3):116-21. doi: 10.3109/0167482X.2013.824418. PMID 23952169
- [Result] Narendran S, Nagarathna R, Narendran V, Gunasheela S, Nagendra HR. Efficacy of yoga on pregnancy outcome. J Altern Complement Med. 2005 Apr;11(2):237-44. doi: 10.1089/acm.2005.11.237. PMID 15865489
- [Result] Jiang Q, Wu Z, Zhou L, Dunlop J, Chen P. Effects of yoga intervention during pregnancy: a review for current status. Am J Perinatol. 2015 May;32(6):503-14. doi: 10.1055/s-0034-1396701. Epub 2014 Dec 23. PMID 25535930
- [Result] Cramer H, Frawley J, Steel A, Hall H, Adams J, Broom A, Sibbritt D. Characteristics of women who practice yoga in different locations during pregnancy. BMJ Open. 2015 Aug 21;5(8):e008641. doi: 10.1136/bmjopen-2015-008641. PMID 26297372
- [Result] Sharma M, Branscum P. Yoga interventions in pregnancy: a qualitative review. J Altern Complement Med. 2015 Apr;21(4):208-16. doi: 10.1089/acm.2014.0033. Epub 2015 Feb 24. PMID 25710094
- [Result] Esencan TY, Karabulut Ö, Yıldırım AD, Abbasoğlu DE, Külek H. et. al. Type of delivery, time of ınitial breastfeeding, and skin-to-skin contact of pregnant women participating in childbirth preparation education. Florence Nightingale Journal of Nursing 2018; 26(1), 31-43. https://doi.org/10.26650/FNJN.387192.
- [Result] Kjergaard H, Wijma K, Dykes AK, Alehagen S. Fear of childbirth in obstetrically low-risk nulliparous women in Sweden and Denmark. Journal of Reproductive and Infant Psychology 2008; 26(4): 340-50.
- See also: Akarsu RH. The effect of pregnancy yoga on the psychosocial health level of pregnant women and prenatal attachment [PhD dissertation],. T.C. Istanbul University, Institute of Health Sciences, Department of Women's Health and Diseases Nursing, Women — http://tez.yok.gov.tr/UlusalTezMerkezi/tezSorguSonucYeni.jsp
- See also: Esencan TY, Karabulut Ö, Yıldırım AD, Abbasoğlu DE, Külek H. et. al. Type of delivery, time of ınitial breastfeeding, and skin-to-skin contact of pregnant women participating in childbirth preparation education. Florence Nightingale Journal of Nursi — http://fnjn.org/en/type-of-delivery-time-of-initial-breastfeeding-and-skin-to-skin-contact-of-pregnant-women-participating-in-childbirth-preparation-education-13668
- Available data/document: PhD thesis — http://tez.yok.gov.tr/UlusalTezMerkezi/tezSorguSonucYeni.jsp

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Randomised (n=115)
  Excluded (n=38):
  Not meeting inclusion criteria (n=30.) Declined to participate (n=8)
Period: Overall Study
Arm/Group | The Study Group | Control Group
Started | 46 | 69
Completed | 30 | 60
Not Completed | 16 | 9
Not completed — Not attending regular yoga class | 16 | 0
Not completed — Not attending the pregnancy school | 0 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | The Study Group | Control Group | Total
Number analyzed (Participants) | 30 | 60 | 90
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 60 | 90
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Standard Deviation); unit: years] | 29.7 (3.44) | 30.2 (4.09) | 29.9 (3.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 60 | 90
  Male | 0 | 0 | 0
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg / m2] | 25.77 (3.26) | 27.37 (4.62) | 26.357 (3.94)

OUTCOME MEASURES:

1. Primary Outcome: Characteristics of Labor (Pregnant)
Description: The Introductory Information Form, which consisted of 8 questions (socio-demographic data) and pregnancy characteristics (12 questions) of pregnant women, and which was prepared in line with the sources, was used.
Time Frame: 16 hours
Measure: Number; unit: participants
Arm/Group | The Study Group | Control Group
Number analyzed (Participants) | 30 | 60
participants
  Electronic Fetal Monitoring | 30 | 59
  Vaginal Examination | 30 | 59
  Movement limitation | 5 | 28
  Enema | 17 | 49
  Induction | 9 | 50
  Normal birth | 24 | 39
  Caesarian | 6 | 21

2. Primary Outcome: Comparison of Visual Analog Scale (Pain) Scores of Pregnant Women in Study and Control Group
Description: The Visual Analog Scale (VAS) consists of a line, often 10 cm long, with verbal anchors at either end, (e.g.,"no pain" on the far left and "the most intense pain imaginable" on the far right). The scale takes a minimum of 0 and a maximum of 10, and higher scores mean a worse result. Visual Analogue Scale (VAS) was used to assess the pains during the birth process of the pregnant women in both the study and control groups.Two ends of the parameter to be evaluated at the two ends of a 100 mm line in VAS the definition is written and the pregnant woman is asked to indicate on this line where her condition is appropriate by drawing a line or putting a dot or pointing. For example, I have no pain at all at one end for pain, very severe pain is written on the other end, and the patient marks his current state on this line. The length of the distance from the place where there is no pain to the place marked by the patient indicates the patient's pain.
Time Frame: the 4th hour on average after the birth
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | The Study Group | Control Group
Number analyzed (Participants) | 30 | 60
units on a scale
  VAS LATENT (This is when pregnant woman cervix becomes soft and thin) | 3.00 (1.84) | 5.48 (1.51)
  VAS ACTIVE (During active labor, cervix will dilate from 4 centimeters (cm) to 7 cm.) | 6.90 (1.88) | 8.80 (0.98)
  VAS TRANSITION (cervix will dilate from 7 to its final 10 centimeters.) | 8.24 (2.12) | 9.86 (0.41)

3. Secondary Outcome: Comparison of WIJMAA and WIJMAB Average Scores of Pregnant Women in the Study and Control Groups
Description: the WIJMA Delivery Expectancy/Experience Questionnaire A, was applied once during the study after the 28th week of pregnancy in preparation for childbirth. Wijma Delivery Expectancy/Experience Questionnaire Version B (W-DEQ B) and was applied in the 4th hour on average after the birth event.W-DEQ A: responses on the 33-point scale numbered from 0 to 5 it is a six-bit likert-type scale. 0 is expressed as" completely "and 5 as" never". The minimum score that can be taken from the scale is 0, while the maximum score is 165. High scores indicate that the fear of childbirth experienced by women is high.W-DEQ B: the scale consists of 32 substances. In scale responses are numbered from 0 to 5 and are of six likert type. 0 is expressed as" completely "and 5 as" never". The minimum score on the scale is 0, while the maximum score is 160. As the score increases, the fear of childbirth experienced by women increases.
Time Frame: the 4th hour on average after the birth
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | The Study Group | Control Group
Number analyzed (Participants) | 30 | 60
score on a scale
  WIJMAA | 47.67 (26.37) | 57.75 (33.27)
  WIJMAB | 29.70 (17.51) | 72.38 (27.32)

4. Secondary Outcome: Comparison of Average Self-sufficiency Scores of Pregnant Women in the Study and Control Groups
Description: The Childbirth Self-Efficacy Scale Short Form was applied twice as the short form to the study and control group during the study. After the start of birth preparation training, when the pregnant women were in the 28th week, after the application of other forms, it was applied as a pre-test and as a post-test at a time when the pregnant women were appropriate. The lowest score, which can be obtained from the lower dimensions of the scale, is 32, and the highest score is 320 points. A high score to be taken from each lower dimension is related to the birth of pregnant women it shows that the expectation of qualification and results is high. As the scores rise it is determined that it increases self-sufficiency.
Time Frame: the 4th hour on average after the birth
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | The Study Group | Control Group
Number analyzed (Participants) | 30 | 60
score on a scale
  Result expectation I | 137.23 (20.21) | 124.32 (27.20)
  Self-sufficiency I | 223.03 (36.83) | 205.80 (40.94)
  Result expectation II | 148.30 (14.10) | 125.30 (19.66)
  Sufficiency expectation II | 139.87 (16.88) | 109.20 (16.91)
  Self-sufficiency II | 288.17 (28.25) | 234.50 (32.00)
Statistical Analysis 1: Comparison: The Study Group vs Control Group; Test type: Superiority — the t-test in independent groups; p < 0.05, t-test, 2 sided; Mean Difference (Net) = 0.02, Standard Deviation 0.80

ADVERSE EVENTS:
Time Frame: Between the 28th week of pregnancy and the 4th hour after birth
Arm/Group | The Study Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/60
Other Adverse Events (participants affected / at risk) | 0/30 | 0/60

LIMITATIONS AND CAVEATS:
The study's being conducted on pregnant women admitted to a training and research hospital on the Anatolian side of Istanbul, high education levels of the pregnant women, and the fact that the participants were determined only in this group were among the limitations of the study. In addition, the results of the study cannot be generalized to the entire population because it was conducted with pregnant women who were healthy and it was their first birth.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No